CLINICAL TRIAL: NCT07269288
Title: Study Protocol on the Correlation and Mechanistic Study of GGCX Gene With Prognosis in Acute Ischemic Stroke
Brief Title: The Correlation and Mechanistic Study of GGCX Gene With Prognosis in Acute Ischemic Stroke
Status: Not yet recruiting | Type: Observational
Sponsor: Peking University Aerospace Center Hospital (Other)
Responsible Party: Principal Investigator, Xia Zhang, Researcher, Aerospace Center Hospital
Other Study IDs: 2025017; 2024PSPT0905100 (Other Grant/Funding Number: NHC-Million Disability Reduction Expert Committee)
Record Dates: First submitted 2025-11-25; First posted 2025-12-08 (Actual); Last update posted 2025-12-08 (Actual); Status verified 2025-11

CONDITIONS: Acute Ischemic Stroke
Keywords: Stroke
MeSH Terms: conditions — Ischemic Stroke; Stroke | interventions — Clinical Protocols

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Acute Ischemic Stroke Group: These subjects were acute ischemic stroke patients who had been followed up for 3-12 months after discharge.
  Interventions: Combination Product: Usually, all enrolled patients with acute ischemic stroke will receive routine medication and/or surgical treatment according to clinical diagnosis and treatment protocols.

INTERVENTIONS:
Combination Product: Usually, all enrolled patients with acute ischemic stroke will receive routine medication and/or surgical treatment according to clinical diagnosis and treatment protocols. — The conventional drug therapy includes anticoagulant, antiplatelet, antihypertensive and other drugs. The surgical therapy includes AIS intravenous thrombolysis or endovascular therapy.

SUMMARY:
This observational study aims to investigate the impact of GGCX gene mutations and GGCX levels on stroke prognosis in patients with ischemic stroke, as well as their correlation. The main issues are:

What is the relationship and potential mechanism between GGCX gene mutations and their expression levels and the composite prognosis of recurrence, death, and bleeding events in patients with ischemic stroke? Collect blood samples from enrolled ischemic stroke patients for genetic testing, and conduct follow-up visits at 3, 6, and 12 months after discharge to evaluate clinical prognosis outcomes. This will answer questions about the relationship and mechanism between GGCX gene and patient prognosis.

ELIGIBILITY:
* Inclusion Criteria

  (1) Inclusion Criteria for Acute Ischemic Stroke Patients:
  1. Aged between 18 and 85 years.
  2. Diagnosed with ischemic stroke (in accordance with the "Chinese Guidelines for Diagnosis and Treatment of Acute Ischemic Stroke 2023," including TOAST etiological/pathogenic subtypes: large-artery atherosclerosis (LAA), cardioembolism (CE), small-artery occlusion (SAO), stroke of other determined etiology (SOE), and stroke of undetermined etiology (SUE)).
  3. Acute onset, with symptoms occurring within 72 hours and being the first episode.
  4. Voluntary participation with signed informed consent.

  (2) Inclusion Criteria for Healthy Controls: 1) Healthy control population matched for age, gender, and risk factors (including personal and family history).
* Exclusion Criteria

  (1) Exclusion Criteria for Healthy Controls:
  1. Patients with cerebrovascular diseases occurring within 72 hours.
  2. Pregnant or lactating patients.

  (2) Exclusion Criteria for Acute Ischemic Stroke Patients:
  1. Other types of stroke, including hemorrhagic stroke, mixed stroke, and tumor-related stroke patients.
  2. Patients with coagulation disorders or other hematologic diseases.
  3. Patients with severe cardiovascular, pulmonary, or hepatic diseases.
  4. Renal dysfunction.
  5. Cancer patients.
  6. Patients with active gastric ulcers or gastric bleeding.
  7. Pregnant or lactating patients.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: This study will be conducted in six hospitals (centers) across the country, namely Xi'an Jiaotong University First Affiliated Hospital, Shandong Weifang Second People's Hospital, Shandong Linshu People's Hospital, Hunan Second People's Hospital (Hunan Brain Hospital), and Nantong First People's Hospital.
Sampling Method: Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2026-01-25 (Estimated); Primary Completion 2026-08-31 (Estimated); Study Completion 2028-02-28 (Estimated)

PRIMARY OUTCOMES:
Evaluate the recurrence, death, and bleeding events of stroke in the research subjects | Follow up will be conducted at 3 months, 6 months, and 12 months after the patient's discharge, and the main outcome events mentioned above will be evaluated.
  Including recurrent ischemic stroke events; Death events include hemorrhagic death, vascular death, and acute myocardial infarction events; Intracranial or other bleeding events (refer to the International Classification of Bleeding Events ICD-10 code).

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University Aerospace Center Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: Undecided
IPD will decide whether to share based on laws and regulations and the management measures of the Clinical Trial Ethics Committee.